CLINICAL TRIAL: NCT02958150
Title: Randomised Clinical Trial: Dexmedetomidine Versus Standard Clinical Practice During Non Invasive Mechanical Ventilation
Brief Title: Dexmedetomidine Versus Standard Clinical Practice During Non Invasive Mechanical Ventilation
Acronym: DEX-PCH-VMNI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Ana Vallejo de la Cueva, Registered Doctor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX-PCH-VMNI
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine according to the stablished protocol
  Interventions: Drug: Dexmedetomidine
- Standard Clinical Practice (Active Comparator): The physician in charge will decide the treatment to be administered (if deemed necessary) in accordance with the protocol established at the department
  Interventions: Procedure: Standard Clinical Practice

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine
Procedure: Standard Clinical Practice
  Arms: Standard Clinical Practice

SUMMARY:
This study compare the effectiveness of dexmedetomidine as a sedative drug during NIV and the different strategies routinely used in patients with ARF of different aetiologies. Efficacy will be assessed based on absence of intubation, short term prognosis, and occurrence of medical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Competent or with legal representative able to sign inform consent.
* Reversible ARF secondary to heart failure, COPD exacerbation, pneumonia, or at risk of pot-extubation failure* who meet the criteria for starting NIV.
* Signs and symptoms of respiratory distress or
* Moderate to severe dyspnoea, grater than usual and/or
* Respiratory rate greater than 25 in COPD or greater than 30 in hypoxemic ARF and/or
* Use of accessory muscles and/or paradoxical breathing and/or
* Hypercapnic encephalopathy
* And changes in gas exchange
* PaCO2>45 mmHg, pH<7.35 and/or
* PaO2/FiO2 between 300 and 150.

  *Patients at risk of post-extubation failure: Patients who meet at least one of the following criteria.
* Impaired consciousness.
* Age over 65 years
* Heart failure with EF >30%
* Severe disease with an Acute Physiology and Chronic Health Evaluation (APSCHE) score >12.
* Protracted weaning before extubation

Exclusion Criteria:

* Respiratory arrest, direct indication of OTI and IMV.
* Severe unstable comorbidity (myocardial ischemia with ejection fraction <30%, arrythmia, uncontrolled hypotension defined as systolic blood pressure less than 90 mmHg with doses of norepinephrine>0.5 mcg/kg/min and/or dobutamine>10 mcg/kg/min).
* Inability to protect the airway: bronchial aspiration.
* Fixed upper airway obstruction.
* Tracheostomy.
* Undrained pneumothorax.
* Severe agitation or lack of collaboration of the patient despite medication administered.
* Facial burns or trauma.
* Facial surgery or anatomical changes which prevent mask fitting.
* Hypersensitivity to the active substance or to any of the excipients listed in section 6.1.
* Allergy to eggs, soya, or peanuts.
* HR< 50 bpm not induced by beta- blockers.
* Advanced heart block (grade 2 or 3) unless paced.
* Acute cerebrovascular conditions.
* Increased intracranial pressure.
* Closed angle glaucoma.
* Myasthenia gravis.
* Concurrent use of CYP3A4 inhibitors (amprenavir, atazanavir, or ritonavir).
* Refuse to participate in the trial.
* Pregnant or nursing patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2022-03 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To determinate the percentage of orotracheal intubations, and thus the need for NIV during the trial. | 72 hours
  Need for intubation is defined as the presence of any of the following: SpO2<80% or P aO2/FiO2<150, seizures, poor secretion management, hypercapnia and pH<7.20, hypotension: systolic blood pressure (SBP)<80 mmHg refractory despite administration of vasoactive amines or electrocardiogram (ECG) with ischaemic changes or ventricular arrhythmia resulting from myocardial hypoxia.

SECONDARY OUTCOMES:
To determinate NIV duration of NIV in each group. | 72 hours
  Number of hours the patient will be on NIV.
To analyse stay at the ICU in each group. | An average of 5 days
  Number of days patients stay at the ICU until they are discharged home or die.
To analyse hospital stay in each group | 15 days
  Number of days patients remain at the hospital until they are discharged home or die.
To compare all-cause mortality at the ICU in both groups. | Through study completion, an average of 3 years
  Percentage of all deaths from any cause in patients with ARF on NIV at the ICU in both study groups.
To compare specific mortality at the ICU in both groups. | Through study completion, an average of 3 years
  Percentage of deaths attributable to ARF in patients on NIV at the ICU in both study groups.
To analyse hospital-specific mortality. | Through study completion, an average of 3 years
  Percentage of all deaths attributable to ARF in patients on NIV at the ICU discharged to a ward in the 2 study groups.
To analyse all-cause hospital mortality. | Through study completion, an average of 3 years
  Percentage of all deaths from any aetiology of ARF in patients treated with NIV in the ICU discharged to a ward in the 2 study groups.
To report the course of ARF in each group. | 1 and 24 hours after NIV
  Based on the presence before the start of NIV
To report NIV tolerance during administration of dexmedetomidine versus SCP. | During administration of dexmedetomidine/SCP and up to 24 hours after drug infusion/SCP is completed.
  Nausea and/or vomiting, Aspiration pneumonia, delirium, agitation, interface tolerance or pain secondary to use of interface.
To report the adverse effects of dexmedetomidine. | During drug administration and up to 24 hours after drug infusion is completed.
  Bradycardia, hypotension, tachycardia, hypertension and/or transient respiratory depression.
To asses patient satisfaction with dexmedetomidine as compared to SCP | Through study completion, an average of 3 years
  Patient satisfaction with use of dexmedetomidine as compared to drugs used in SCP will be estimated once NIV and dexmedetomidine/SCP infusion have been completed, using a Likert type questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Vallejo, Principal Investigator — Basque Health Service: Araba University Hospital
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Álava, Spain